CLINICAL TRIAL: NCT04443023
Title: Randomized Comparison of Eligible TAVI-valves - Cohort B (Sapien Versus Myval)
Brief Title: Comparison of Eligible TAVI-valves - Cohort B
Acronym: Compare-TAVI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Odense University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Christian Juhl Terkelsen, Principal investigator, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Compare-TAVI
Record Dates: First submitted 2020-06-07; First posted 2020-06-23 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Transcatheter Aortic Valve Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sapien (Active Comparator): Patients randomized to treatment
  Interventions: Device: chosen TAVI valve
- Myval (Active Comparator): Patients randomized to treatment
  Interventions: Device: chosen TAVI valve

INTERVENTIONS:
Device: chosen TAVI valve — chosen TAVI valve

SUMMARY:
The study performs head-to-head comparison of two TAVI-valves: Sapien and Myval.

DETAILED DESCRIPTION:
The purpose of the present study is to ensure a continuous comparison of the TAVI-valves implanted, and to monitor long-term valve performances.

Purpose: To randomize between two TAVI-valve types in patients who according to a heart team conference is found eligible for treatment with more than one valve.

Hypotheses:

1. There is no difference in the combined endpoint (death, stroke, moderate/severe para-valvular leakage, moderate/severe device stenosis) between the two valves to be compared.
2. There is no difference between valves in secondary endpoints: death, stroke, moderate/major paravalvular leakage, moderate/severe aortic device stenosis, new pacemaker implantation, readmission for congestive heart failure, 6-minute walk test, and degeneration of the valve as evaluated by computerized tomography (HCT), transthoracic echocardiography (TTE), transesophageal echocardiography (TEE), or MRI.

Design: Randomized controlled trial with clinical national registry follow-up.

Centers eligible for inclusion: Scandinavian and European centers who fulfill the above mentioned criteria.

Randomization:

Before randomizing patients, the center decides which two valves the patient is found eligible for, and enters these valves in the electronic randomization form (TrialPartner). Randomization is then performed between these two valves. A patient is only randomized if a dedicated technical TAVI conference has found the patient eligible for treatment with both valves.

Consecutive cohorts are established.

In the current study we plan to initiate the following cohorts:

Cohort B: Patients randomized to the Sapien or the Myval TAVI valve.

Operator requirements:

Any procedure requires that the physician has performed at least 15 implantations with the valve in use. Otherwise the procedure is performed according to the routine of the institution.

ELIGIBILITY:
Inclusion Criteria:

1. Patient more than 18 years of age.
2. Patient eligible for at least 2 valves being implanted routinely at the participating center, according to a TAVI heart team conference.
3. The center experience for each of the valves considered should be more than 15 cases a year, and at least 15 valves implanted before a valve can be used in the trial.
4. The center volume should be more than 75 cases a year.
5. The patient has given signed informed consent.
6. TAVI performed via the femoral artery.

Exclusion Criteria:

1. Not able to give written inform consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1031 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2034-11-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with MACE (Major Adverse Cardiovascular Events) | 1 year
  Mortality, stroke, moderate/major PVL, moderate/severe aortic device stenosis at 1 year, using VARC-3 criteria

SECONDARY OUTCOMES:
Percentage of patients with MACE | 30 day, 3-year, 5-year and 10-year
  Mortality, stroke, moderate/major paravalvular leakage (PVL), moderate/severe aortic device stenosis at 1 year, using VARC-3 criteria
Percentage death | 30-day, 1-year, 3-year, 5-year, 10-year
  Mortality
Percentage of patients with stroke | During admission, 30-day, 1-year, 3-year, 5-year, 10-year
  According to Valve Academic Research Consortium (VARC)-3 criteria
Percentage of patients with moderate or severe paravalvular leakage | 30-day, 1-year, 3-year, 5-year, 10-year
  Moderate or severe paravalvular leakage according to VARC-3 criteria
Percentage of patients with moderate/major aortic stenosis | 30-day, 1-year, 3-year, 5-year, 10-year
  According to VARC-3 criteria
Percentage of patients with new pacemaker | During admission, 30-day, 1-year, 3-year, 5-year, 10-year
  New Pacemaker after TAVI-procedure
Percentage of patients with major bleeding | 30-day, 1-year, 3-year, 5-year, 10-year
  Major bleeding according to Bleeding Academic Research Consortium (BARC) type 3 or 5 criteria, resulting in either a drop in Hbg>=1.86 mmol/l or >=2 units of blood transfusion
Distance in meters during 6-minute walk test | 30-day, 1-year, 3-year, 5-year, 10-year
  6-minute walk test
Percentage of patients with other TAVI-related complications | During TAVI-procedure
  conversion to open surgery during implantation, unplanned use of cardiopulmonary support (CPS), coronary artery obstruction, ventricular septal perforation, mitral valve apparatus damage or dysfunction, cardiac tamponade, valve thrombosis, valve embolization, valve migration, need for TAVI-in-TAVI deployment, using VARC-3 criteria
Percentage of patients with endocarditis | 30-day, 1-year, 3-year, 5-year, 10-year
  Endocarditis
Proportion with successful implantation of the chosen valve. | During procedure
  This means no need for more than 1 TAVI valve, no change to another valve than planned during the procedure because it was impossible to implant the valve planned, and no conversion to surgery or procedure-related death.
Percentage of patients with major vascular access site and access-related complications | During admission and 30-day
  According to VARC-3 criteria
Percentage of patients with valve thrombosis or severe stenosis | 30-day, 1-year, 3-year, 5-year, 10-year
  Valve thrombosis or severe stenosis confirmed by Echo or HCT
Percentage of patients with readmission with congestive heart failure | 30-day, 1-year, 3-year, 5-year, 10-year
  Readmission with congestive heart failure
Percentage of patients with increase in creatinin level of 100% or more, or dialysis | during admission and within 30 days
  Increase in renal creatinine level more than to >=200% (AKIN stage 2-3, VARC-3 criteria) or dialysis
Percentage of patients with moderate/severe PVL stratified according to level of annular calcium on HCT in three groups | 30-day
  Severity of PVL stratified according to level of annular calcium on HCT (low/medium/high)
Mean Gradient (AO) stratified according to level of annular calcium on HCT in three groups | 30-day
  Gradient (AO) stratified according to level of annular calcium on HCT (low/medium/high)
Percentage of patients with prosthesis-patient mismatch | 30-day, 1-year, 3-year, 5-year, 10-year
  Prosthesis-patient mismatch (EOA/body surface area). Severe PPM≤0.65 cm2/m2. Moderate PPM≤0.85 cm2/m2 according to VARC-3 criteria
Mean effective orifice area measured by MRI | 30-day
  Effective orifice area measured by MRI in patients participating in MRI-substudy
Percentage of patients with leaflet thickening (hypoattenuated leaflet thickening = HALT) or reduced leaflet motion or thrombus assessed by HCT | 30-day and 1-year
  Leaflet thickening (hypoattenuated leaflet thickening = HALT) or reduced leaflet motion or thrombus assessed by HCT in patients participating in HCT-substudy
Mean volume of aortic regurgitation measured by MRI | 30-day
  Volume of aortic regurgitation measured by MRI in patients participating in MRI-substudy
Other tavi-related complications | 30-day
  Anulus rupture or aortic rupture
AMI | 30-day, 1-year, 3-year, 5-year and 10-year
  Acute Myocardial Infarction
PCI og CABG | 30-day, 1-year, 3-year, 5-year and 10-year
  Percutaneous Coronary Intervention or coronary artery bypass grafting
Reopeation | 30-day, 1-year, 3-year, 5-year and 10-year
  Reopeation with TAVI, Surgical ortic valve replacement (SAVR) or BAV (Balloon aortic valvuloplasty) according to VARC-3 criteria
Afib | 30-day, 1-year, 3-year, 5-year and 10-year.
  Newly diagnosed atrial fibrillation according to VARC-3 criteria

CONTACTS AND LOCATIONS:
Overall Officials: henrik nissen, PhD, Study Chair — odense univeristy hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Normally this will be possible when data are published and anonymized. Mainly to support meta-analysis on individual level data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When endpoints are published in an international peer-reviewed paper
Access Criteria: To share data there shall be a well-defined purpose. This could be to contribute to a meta-analysis on individual level data.

REFERENCES:
- [Background] Terkelsen CJ, Thim T, Freeman P, Dahl JS, Norgaard BL, Kim WY, Tang M, Sorensen HT, Christiansen EH, Nissen H. Randomized comparison of TAVI valves: The Compare-TAVI trial. Am Heart J. 2024 Aug;274:84-94. doi: 10.1016/j.ahj.2024.05.003. Epub 2024 May 9. PMID 38729550
- [Derived] Terkelsen CJ, Freeman P, Dahl JS, Thim T, Norgaard BL, Mogensen NSB, Tang M, Eftekhari A, Povlsen JA, Poulsen SH, Pedersen L, Hjort J, Ellert J, Christiansen EH, Sorensen HT, Nissen H. SAPIEN 3 versus Myval transcatheter heart valves for transcatheter aortic valve implantation (COMPARE-TAVI 1): a multicentre, randomised, non-inferiority trial. Lancet. 2025 Apr 19;405(10487):1362-1372. doi: 10.1016/S0140-6736(25)00106-0. Epub 2025 Apr 2. PMID 40187364

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Original protocol (2023-05-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT04443023/Prot_SAP_000.pdf